CLINICAL TRIAL: NCT04668378
Title: Effects of Time-restricted Eating and Resistance Training on Body Composition, Inflammatory Markers and Cardiometabolic Risk Factors
Brief Title: Effects of a Time Restricted Eating Protocol on Resistance Training Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Antonio Paoli, Full Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TRE-RET
Record Dates: First submitted 2020-12-04; First posted 2020-12-16 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Fasting; Healthy
Keywords: fasting; time restricted eating; resistance training; body composition; inflammation
MeSH Terms: conditions — Fasting; Intermittent Fasting; Inflammation

STUDY DESIGN:
Intervention Model Description: It is a single blind, parallel arms study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Time restricted eating (TRE) - two month (Experimental): partecipants underwent 2 months of a TRE protocol, during which they consumed 100% of the daily energy needs in an 8-hour time window: from 1:00 PM to 8:00 PM. Body composition, muscle strength and blood parameters were measured before and after the diet intervention.
  Interventions: Other: Time restricted eating
- Normal Diet (ND) - two month (Active Comparator): partecipants underwent 2 months of a regular diet schedule and consumed 100% of the daily energy needs in 3 meals between 8:00 AM and 8:00 PM. Body composition, muscle strength and blood parameters were measured before and after the diet intervention.
  Interventions: Other: Normal Diet
- Time restricted eating (TRE) - twelve month (Experimental): partecipants underwent 12 months of a TRE protocol, during which they consumed 100% of the daily energy needs in an 8-hour time window: from 1:00 PM to 8:00 PM. Body composition, muscle strength and blood parameters were measured before and after the diet intervention.
  Interventions: Other: Time restricted eating
- Normal Diet (ND) - twelve month (Active Comparator): partecipants underwent 12 months of a regular diet schedule and consumed 100% of the daily energy needs in 3 meals between 8:00 AM and 8:00 PM. Body composition, muscle strength and blood parameters were measured before and after the diet intervention.
  Interventions: Other: Normal Diet

INTERVENTIONS:
Other: Time restricted eating — TRE subjects consumed 100 % of their energy needs divided into three meals consumed at 1 p.m., 4 p.m. and 8 p.m., and fasted for the remaining 16 h per 24-h period.
  Arms: Time restricted eating (TRE) - twelve month; Time restricted eating (TRE) - two month
Other: Normal Diet — ND group ingested their caloric intake as three meals consumed at 8 a.m., 1 p.m. and 8 p.m.
  Arms: Normal Diet (ND) - twelve month; Normal Diet (ND) - two month

SUMMARY:
The study sought to investigate the effects of 16/8 time restricted eating (TRE) with windows of 16 hours of fasting and 8 hours of eating on on body composition, muscle strength, and metabolic factors during resistance training in healthy resistance trained males

DETAILED DESCRIPTION:
Thirty-four resistance-trained males were randomly assigned to a TRE group or to a control normal pattern group (ND) with a traditional meal pattern. The TRE group consumed 100% of the daily energy needs in an 8-hour time window: from 1PM (post meridiem) to 8:00 PM whilst the ND group consumed 100% of their daily energy needs in 3 meals between 8:00 AM (ante meridiem) and 8:00 PM. During the experimental period, training loads were similar and standardize in the two groups. partecipants were tested before and after 8 weeks of the intervention. Body composition , basal metabolism, performances indexes and blood parameters were measured. After the completition of the first two months of study, subjects were ask to volunteer to continue the intervention for 10 extra months. A total of twenty subjects from, 10 from each group (TRE or ND) continued and completed the second part of the study.

ELIGIBILITY:
Inclusion Criteria:

* continuously engaged in resistance training for at least 5 years
* at least 3 years experience in split training routines
* male

Exclusion Criteria:

* adherence to special diets
* use of nutritional supplements (except a daily multivitamin-mineral and/or protein supplement)
* use of steroids
* use of medications

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Fat Mass | change from baseline to up to 2 months
  fat mass measured dual energy X-ray absorptiometry (DXA)
Fat Free Mass | change from baseline to up to 2 months
  fat free mass measured dual energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Fat Mass | change from baseline to up to 12 months
  fat mass measured dual energy X-ray absorptiometry (DXA)
Fat Free Mass | change from baseline to up to 12 months
  fat free mass measured dual energy X-ray absorptiometry (DXA)
total cholesterol | change from baseline to up to 2 months
  total cholesterol as milligram per deciliter
total cholesterol | change from baseline to up to 12 months
  total cholesterol as milligram per deciliter
glucose | change from baseline to up to 2 months
  glucose as milligram per deciliter
glucose | change from baseline to up to 12 months
  glucose as milligram per deciliter
Leg muscle strength | change from baseline to up to 2 months
  Leg muscle strength measured via via 1-RM test
Leg muscle strength | change from baseline to up to 12 months
  Leg muscle strength measured via via 1-RM test

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paoli, MD, Principal Investigator — University of Padova
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moro T, Tinsley G, Pacelli FQ, Marcolin G, Bianco A, Paoli A. Twelve Months of Time-restricted Eating and Resistance Training Improves Inflammatory Markers and Cardiometabolic Risk Factors. Med Sci Sports Exerc. 2021 Dec 1;53(12):2577-2585. doi: 10.1249/MSS.0000000000002738. PMID 34649266